CLINICAL TRIAL: NCT06835413
Title: Monitoring Combined Effect of Balance and Strengthening Exercises on Static and Dynamic Balance in Elderly Populations
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: South Valley University (Other)
Responsible Party: Principal Investigator, Ibrahim Abuzaid, Head of Department of physical therapy for cardiovascular/pulmonary disorders and Geriatrics, South Valley University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: South Valley University PT
Record Dates: First submitted 2025-02-08; First posted 2025-02-19 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2025-02

CONDITIONS: Geriatrics Balance Disturbance With High Risk Falling, Osteoporosis, Vestibular Age Related Changes, Female Post-menopausal Based on History
Keywords: 1-Static balance; 2- dynamic balance; 3- Geriatrics populations; 4- Balance exercises; 5-Strengthening exercises
MeSH Terms: conditions — Osteoporosis

STUDY DESIGN:
Intervention Model Description: The study Group: training program will be implemented for 60 min per session, 3 times per week for 8 weeks. This intervention included aerobic training on treadmill or bicycle ergometer and mat activities (stretching and muscle strengthening). Balance Exercises & Strength and Balance Exercises.
  1-Balance Exercises A- Standing with a decreased base B- Graded reaching in standing C- Stepping in different directions D- Walking practice A- Standing with a decreased base B- Graded reaching in standing
  * Feet together and level.
  * Semi-tandem stance.
  * Tandem stance.
  * Stand on one leg.
  * Maintain position for longer
  * Close eyes.
  * Stand on different surfaces e.g. foam rubber mat.
  * Minimize hand support & Aim to increase time without hand support. • Feet placement- narrower, step standing
  * Reaching further.
  * Reaching in different directions.
  * Reaching down to a stool or the floor.
  * Reaching for heavier objects.
  * Reaching for a full cup of water.
  * Standing on a softer surface eg foam
Who Masked: Participant
Masking Description: The study Group: training program will be implemented for 60 min per session, 3 times per week for 8 weeks. This intervention included aerobic training on treadmill or bicycle ergometer and mat activities (stretching and muscle strengthening). Balance Exercises & Strength and Balance Exercises.
  1-Balance Exercises A- Standing with a decreased base B- Graded reaching in standing C- Stepping in different directions D- Walking practice A- Standing with a decreased base B- Graded reaching in standing
  * Feet together and level.
  * Semi-tandem stance.
  * Tandem stance.
  * Stand on one leg.
  * Maintain position for longer
  * Close eyes.
  * Stand on different surfaces e.g. foam rubber mat.
  * Minimize hand support & Aim to increase time without hand support. • Feet placement- narrower, step standing
  * Reaching further.
  * Reaching in different directions.
  * Reaching down to a stool or the floor.
  * Reaching for heavier objects.
  * Reaching for a full cup of water.
  * Standing on a softer surface eg foam
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The study Group (Experimental): training program will be implemented for 60 min per session, 3 times per week for 8 weeks. This intervention included aerobic training on treadmill or bicycle ergometer and mat activities (stretching and muscle strengthening). Balance Exercises & Strength and Balance Exercises.
  1. Balance Exercises A- Standing with a decreased base B- Graded reaching in standing C- Stepping in different directions D- Walking practice
  2. Strength and Balance Exercises A- Sit-to-stand B- Heel raise C- Forward step-up D- Lateral step-up E- Half- squats sliding down a wall
  Interventions: Procedure: 1-Balance Exercises A- Standing with a decreased base B- Graded reaching in standing C- Stepping in different directions D- Walking practice 2-Strength and Balance Exercises A- Sit-to-stand B- Heel r
- The control group (Active Comparator): The active control group will be received only physical therapy training, which will be provided 3 times per week for 60-min per session. This intervention included aerobic training on treadmill or bicycle ergometer and mat activities (stretching and muscle strengthening).
  Interventions: Procedure: 1-Balance Exercises A- Standing with a decreased base B- Graded reaching in standing C- Stepping in different directions D- Walking practice 2-Strength and Balance Exercises A- Sit-to-stand B- Heel r

INTERVENTIONS:
Procedure: 1-Balance Exercises A- Standing with a decreased base B- Graded reaching in standing C- Stepping in different directions D- Walking practice 2-Strength and Balance Exercises A- Sit-to-stand B- Heel r — 1-Balance Exercises A- Standing with a decreased base B- Graded reaching in standing C- Stepping in different directions D- Walking practice A- Standing with a decreased base B- Graded reaching in standing
  * Feet together and level.
  * Semi-tandem stance.
  * Tandem stance.
  * Stand on one leg.
  * Maintain position for longer
  * Close eyes.
  * Stand on different surfaces e.g. foam rubber mat.
  * Minimize hand support & Aim to increase time without hand support. • Feet placement- narrower, step standing
  * Reaching further.
  * Reaching in different directions.
  * Reaching down to a stool or the floor.
  * Reaching for heavier objects.
  * Reaching for a full cup of water.
  * Standing on a softer surface eg foam rubber mat.
  * Stepping while reaching. C- Stepping in different directions D- Walking Practice
  * Narrow foot position.
  * Longer steps.
  * Faster steps.
  * Step over objects.
  * Choice component e.g. step forward with left foot.
  * Incorporate pivoting on the non-stepping foot.
  * Use different color

SUMMARY:
The purpose of training is to evoke improvements in reactive balance, then the training program may be associated with all postural control systems, including the musculoskeletal system, the cognitive system, as well as the somatosensory feedback system, while challenging the body in different environmental situations and unexpected perturbations

DETAILED DESCRIPTION:
A study will be conducted at South Valley University Hospital. Subjects have been assigned a consent form before enrolling in the study. This study followed the Consolidated Standards of Reporting Trials guidelines.

Design Parallel double blinded randomized control trial. Subjects Study will be included 60 subjects with geriatrics balance disturbance with high risk falling, osteoporosis, vestibular age related changes, female post-menopausal based on history, physical examination. Male and female subjects meeting the following criteria were included: age ranged from 50 to 70 years, BMI was 18-25 kg/m2, will be divided into two groups, If a patient had a history of hiatus hernia, substantial gastro-esophageal reflux, acute cardiac events, un controlled diabetes mellitus, hypertension within the last six weeks, congestive heart failure, acute exacerbation, exacerbation six months before, active hemoptysis, or malignant disease, they were excluded from the study.

Procedures Assessment

Assessment Tools to effectively monitor the combined effects of these exercises, various assessment tools can be employed:

Balance Tests: Standardized tests functional reach and the Timed Up and Go (TUG) test can provide quantitative measures of balance improvements.

* Timed Up and Go (TUG) Method: The patient starts in a seated position. The patient stands up upon therapist's command: walks 3 meters, turns around, walks back to the chair and sits down. The time stops when the patient is seated. The subject is allowed to use an assistive device. Normal time ( < 10 sec)
* Functional Reach Test (FRT): Functional Reach Test is a measure of how high someone can reach while standing. Procedure: If measuring against a wall, the subject stands side on and reaches up with the hand closest to the wall. Keeping the feet flat on the ground, the point of the fingertips is marked then the distance measured. Normal distance 25 centimetres or more (4).

The study Group: training program will be implemented for 60 min per session, 3 times per week for 8 weeks. This intervention included aerobic training on treadmill or bicycle ergometer and mat activities (stretching and muscle strengthening). Balance Exercises & Strength and Balance Exercises.

1. Balance Exercises A- Standing with a decreased base B- Graded reaching in standing C- Stepping in different directions D- Walking practice A- Standing with a decreased base B- Graded reaching in standing

   * Feet together and level.
   * Semi-tandem stance.
   * Tandem stance.
   * Stand on one leg.
   * Maintain position for longer
   * Close eyes.
   * Stand on different surfaces e.g. foam rubber mat.
   * Minimize hand support & Aim to increase time without hand support. • Feet placement- narrower, step standing
   * Reaching further.
   * Reaching in different directions.
   * Reaching down to a stool or the floor.
   * Reaching for heavier objects.
   * Reaching for a full cup of water.
   * Standing on a softer surface eg foam rubber mat.
   * Stepping while reaching. C- Stepping in different directions D- Walking Practice
   * Narrow foot position.
   * Longer steps.
   * Faster steps.
   * Step over objects.
   * Choice component e.g. step forward with left foot.
   * Incorporate pivoting on the non-stepping foot.
   * Use different colors, numbers of letters or a clock face or coins as targets for variety. • Decrease base of support i.e. progress to tandem walk.
   * Increased step size.
   * Increase speed.
   * Change direction.
   * Walk on different surfaces.
   * Walk sideways, backwards.
   * Obstacles to step over and walk around.
2. Strength and Balance Exercises A- Sit-to-stand B- Heel raise C- Forward step-up D- Lateral step-up E- Half- squats sliding down a wall A- Sit-to-stand B- Heel raise

   * Lowering the height.
   * Don't use hands to push off, cross arms across chest.
   * Changing the nature of the surface (e.g. softer chair). • Decrease hand support.
   * Hold the raise for longer.
   * One leg at a time.
   * Adding weight (either vest or belt)
   * Use a wedge to increase the range of motion. C- Forward- Lateral step-up D- Half- squats sliding down a wall
   * Increasing step height.
   * Adding weight (either vest or belt).
   * Decrease hand support.
   * Step up and over block. • Decrease hand support.
   * Hold the squat for longer.
   * Move a short distance away from the wall.
   * Adding weight (either vest or belt).
   * The person can just do 2 sets of 10- 15 repetitions (10-15) repetition maximum (RM).
   * Frequency 3-4 times per week.
   * Intensity of exercise should be limited so that blood pressures not exceed 170 mmHg.
   * Duration of the exercise divided into warm up of 5-10 min, stimulus phase of 30-45 min and cool down of 5 -10 min.

The control group: The active control group will be received only physical therapy training, which will be provided 3 times per week for 60-min per session. This intervention included aerobic training on treadmill or bicycle ergometer and mat activities (stretching and muscle strengthening).

ELIGIBILITY:
Inclusion Criteria:

* geriatrics balance disturbance with high risk falling
* osteoporosis
* vestibular age related changes
* female post-menopausal based on history

Exclusion Criteria:

* Hiatus hernia
* Substantial gastro-esophageal reflux
* Acute cardiac events
* Uncontrolled diabetes mellitus
* Hypertension within the last six weeks
* Congestive heart failure,
* Acute exacerbation, exacerbation six months before
* Active hemoptysis, or malignant disease

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-05-15 (Estimated); Primary Completion 2025-10-15 (Estimated); Study Completion 2026-01-15 (Estimated)

PRIMARY OUTCOMES:
Timed Up and Go (TUG) (sec.) | 8 weeks
  Assessment Tools to effectively monitor the combined effects of these exercises, various assessment tools can be employed:
  • Timed Up and Go (TUG) Method: The patient starts in a seated position. The patient stands up upon therapist's command: walks 3 meters, turns around, walks back to the chair and sits down. The time stops when the patient is seated. The subject is allowed to use an assistive device. Normal time ( < 10 sec)
Functional Reach Test (FRT) (centimeters) | 8 weeks
  Assessment Tools to effectively monitor the combined effects of these exercises, various assessment tools can be employed:
  • Functional Reach Test (FRT): Functional Reach Test is a measure of how high someone can reach while standing. Procedure: If measuring against a wall, the subject stands side on and reaches up with the hand closest to the wall. Keeping the feet flat on the ground, the point of the fingertips is marked then the distance measured. Normal distance 25 centimeters or more

CONTACTS AND LOCATIONS:
Locations (1):
- South Valley university, Qina, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
Undecided

REFERENCES:
- [Result] Bulat T, Hart-Hughes S, Ahmed S, Quigley P, Palacios P, Werner DC, Foulis P. Effect of a group-based exercise program on balance in elderly. Clin Interv Aging. 2007;2(4):655-60. doi: 10.2147/cia.s204. PMID 18225467
- [Result] Hafstrom A, Malmstrom EM, Terden J, Fransson PA, Magnusson M. Improved Balance Confidence and Stability for Elderly After 6 Weeks of a Multimodal Self-Administered Balance-Enhancing Exercise Program: A Randomized Single Arm Crossover Study. Gerontol Geriatr Med. 2016 Apr 26;2:2333721416644149. doi: 10.1177/2333721416644149. eCollection 2016 Jan-Dec. PMID 28138495
- [Result] Zouita S, Zouhal H, Ferchichi H, Paillard T, Dziri C, Hackney AC, Laher I, Granacher U, Ben Moussa Zouita A. Effects of Combined Balance and Strength Training on Measures of Balance and Muscle Strength in Older Women With a History of Falls. Front Physiol. 2020 Dec 23;11:619016. doi: 10.3389/fphys.2020.619016. eCollection 2020. PMID 33424642
- [Result] Dunsky A. The Effect of Balance and Coordination Exercises on Quality of Life in Older Adults: A Mini-Review. Front Aging Neurosci. 2019 Nov 15;11:318. doi: 10.3389/fnagi.2019.00318. eCollection 2019. PMID 31803048
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/31803048/